CLINICAL TRIAL: NCT05821153
Title: Phase I Trial Using Interleukin-2 (IL-2) to Expand Regulatory T Cells in Patients With Alzheimer's Disease
Brief Title: Low Dose IL2 Immunotherapy in AD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Alireza Faridar, Assistant Professor, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00021747
Record Dates: First submitted 2023-03-27; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Aldesleukin — Low dose Interleukin-2 (Aldesleukin) administration to expand Regulatory T cells

SUMMARY:
Neuroinflammation is a significant component of Alzheimer disease (AD). Our data demonstrated compromised regulatory T cells (Tregs) phenotype and suppressive function in AD patients, skewing the immune system toward a proinflammatory status and potentially contributing in disease progression. Low dose interleukin-2 (IL-2) is now viewed as a very promising immunoregulatory drug having the capacity to selectively expand and restore functional Tregs. This study is a phase I open-label study to assess subcutaneous interleukin-2 (IL2) safety and potential efficacy as a Treg inducer in AD. 8 Alzheimer dementia patients with mild clinical dementia will be recruited into the study. The baseline cognitive status will be evaluated in these patients. Monthly five-day-courses of subcutaneous IL2 (1MUI/day) will be administered for a total of 4 months. Changes in Tregs from pre to post injections will be measured during the study period. The expected time participants will be in the study is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer disease according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria13.
* Male or female age 60 to 86 years
* Clinical dementia rating scale of 1
* Total bilirubin less than or equal to 1.5mg/dL
* Alanine aminotransferase level (ALT) less than or equal to five times normal, albumin greater than or equal to 3.0gm/dL
* Serum creatinine less than 1.5 mg/dL
* English language speaking
* A family member or caretaker who is expected to be consistently available, administer study drug and attend study visits throughout the study.

Exclusion Criteria:

* Serious, active bacterial, fungal or viral infection
* Severe pulmonary dysfunction. FEV1 and FVC less than 40% of predicted (or 3 SD below normal) at baseline, If a pulmonary function test is clinically indicated. Hx of intubation for >72 hours.
* Severe cardiac dysfunction defined as left ventricular ejection fraction <40% if an echocardiogram is medically indicated to clarify ongoing symptoms or EKG findings.; a history of non-controlled cardiac arrhythmias; history of cardiac tamponade; Unstable angina or MI in the last 3 months
* Hypersensitivity or allergy to IL-2
* Bowel ischemia/perforation, GI bleeding requiring surgery
* Resistant seizures, history of coma or toxic psychosis lasting >48 hours
* Patients with White Blood Count (WBC) <4,000/mm3; platelets <100,000/mm3; hematocrit (HCT) <30%.

Ages: 60 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
To assess the safety and the tolerability of IL-2 in AD patients | 4 months treatment phase
  Primary endpoints:
  - Number of participants with adverse events and with abnormal laboratory findings (serum chemistry, hematology).

SECONDARY OUTCOMES:
To investigate the impact of low dose IL-2 administration on the blood Treg population in AD patients. | 4 months treatment phase
  Secondary endpoints:
  - Change in Treg percentage out of total # of CD4 cells from baseline to month 4

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Faridar, Principal Investigator — Houston Methodist Neurological Institute
Locations (1):
- Alireza Faridar, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Faridar A, Eid AM, Thome AD, Zhao W, Beers DR, Pascual MB, Nakawah MO, Roman GC, Davis CS, Grundman M, Masdeu JC, Appel SH. A phase 1 open-label pilot study of low-dose interleukine-2 immunotherapy in patients with Alzheimer's disease. Transl Neurodegener. 2023 Nov 16;12(1):54. doi: 10.1186/s40035-023-00387-5. PMID 37968718